CLINICAL TRIAL: NCT03820921
Title: PD-L1 and MMR Status Provided by Endoscopic Ultrasound-Guided Fine-Needle Biopsies as a Predictor of PrognosiS in Patients With Pancreatic Ductal Adenocarcinoma
Brief Title: Evaluation of MMR Status and PD-L1 Expression Using Specimens Obtained by EUS-FNB in Patients With Pancreatic Cancer
Acronym: SUCCESS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ponderas Academic Hospital (Other)
Collaborators: University of Medicine and Pharmacy Craiova (Other)
Responsible Party: Principal Investigator, alina constantin, principal investigator, Ponderas Academic Hospital
Other Study IDs: SUCCESS
Record Dates: First submitted 2018-12-30; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Cancer
Keywords: EUS-FNB, PDL1, MMR
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PATIENTS WITH PANCREATIC CANCER: All patients with a suspicion of pancreatic masses will undergo EUS (including EUS-FNB for confirmation of diagnosis). A positive cytological diagnosis will be taken as a final proof of malignancy of the pancreas mass. The diagnoses obtained by EUS-FNB will be further verified during a clinical follow-up of at least 6 months.
  Immunochemistry will be performed on the EUS-FNB specimens to determine PD-L1 expression and MMR status
  Interventions: Diagnostic Test: EUS-FNB; Other: Immunohistochemistry

INTERVENTIONS:
Diagnostic Test: EUS-FNB — EUS WITH EUS-FNB will be performed for confirmation of diagnosis and analysis of MMR status and PD-L1 expression
  Protocol of EUS with EUS-FNB should include linear EUS instruments with complete examinations of the pancreas. Tumor characteristics (echogenicity, echostructure, size) will be described as well as presence/absence of power Doppler signals.
  EUS-FNB will be performed in all pancreatic masses with at least three passes in the absence of an onsite cytopathologist using a fanning technique with a 22-gauge needle (SharkCore FNB needle Medtronic Corp. or Acquire FNB needle Boston, MA).
Other: Immunohistochemistry — IHC will be performed on treatment-naïve formalin-fixed paraffin-embedded EUS-FNB pancreatic specimens. Briefly, 4-μm-thick tissue sections will be stained using the Ventana BenchMark XT automated slide-staining system using the following antibodies: Anti-PD-L1 (clone SP263, VENTANA, Tucson, AZ), MLH1 (clone G168-728, Cell Marque, Rocklin, California, United States), MSH2 (clone FE11, Biocare Medical, Concord, Massachusetts, United States), MSH6 (clone BC/44, Biocare Medical, Concord, Massachusetts, United States), and PMS2 (clone A16-4, Biocare Medical, Concord, M Massachusetts, United States). Antigen-antibody reactions will be visualized using UltraView detection with diaminobenzidine as the chromogen. The specimen will be considered to have PD-L1 expression if PD-L1 is expressed in ≥ 1 % of tumor cells and a high level of expression if ≥ 50 %. Tumors will be classified as dMMR if they exhibit absent nuclear staining of DNA mismatch repair proteins (MLH1, MSH2, MSH6, or PMS2).

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) has a suboptimal response to standard therapies that modestly impact survival due to its ability to evade host immune surveillance. Emerging evidence has shown that the co-inhibitory receptors, such as programmed death 1 (PD-1), play a critical role in cancer immune-editing. Programmed death-ligand 1 (PD-L1) is an immune checkpoint that is often activated in cancer and plays a pivotal role in the initiation and progression of cancer. The advent of immunotherapy, with checkpoint inhibitors, which block PD-L1 interaction between tumor cells and activated T cells, has significantly altered the treatment algorithm for several solid tumors.

However, the clinicopathologic significance and prognostic value of PD-L1 in PDAC remains controversial. The main technical ground may be that PDAC PD-L1 expression quantification is limited to surgical resection specimens and dependent on specific immunohistochemistry (IHC) tests. In addition, PD-L1 expression has not been extensively assessed before surgery in treatment-naive PDAC patients, due to the current IHC test requirement for a histologic rather than a cytologic evaluation. However, a recent study showed that EUS-fine needle biopsy (FNB) can successfully determine primary pancreas malignancy PD-L1 status.

One recently identified subtype within the genomic landscape of PDAC is the mismatch repair-deficient (dMMR) tumor. Evaluation of dMMR status is particularly important following the FDA approval of the PD-1 inhibitor, pembrolizumab, for the treatment of unresectable or metastatic, microsatellite instability-high (MSI-H) or dMMR PDAC that have progressed following prior treatment, and have no satisfactory alternative treatment options.

The objectives of the project will include the assessment of tumor PD-L1/dMMR expression in patients with PDAC using EUS-FNB samples and the prospective correlation of MMR status and PD-L1 expression with overall survival and progression-free survival of PDAC patients.

ELIGIBILITY:
Inclusion Criteria

* Age 18 to 90 years old
* men or women
* signed informed consent for EUS and EUS -FNB
* the diagnosis of adenocarcinoma histologically confirmed by FNB
* resectable, Unresectable, locally advanced and/or metastatic disease

Exclusion Criteria:

-previous chemotherapy or radiotherapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of pancreatic ductal adenocarcinoma
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of PD-L1 expression analysis on EUS-FNB pancreatic specimens | 1 year
  the percentage of cases where EUS-FNB material was adequate to determine PDL-1 expression
Feasibility of MMR status analysis on EUS-FNB pancreatic specimens | 1 year
  the percentage of cases where EUS-FNB material was adequate to determine MMR status

SECONDARY OUTCOMES:
Tumor response | 3 months
  Tumor response will be assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST). According to RECIST guidelines,complete response (CR) is defined as the complete disappearance of the tumor, partial response (PR) as ≥30% decrease in longest diameter (LD), progressive disease (PD) as ≥20% increase in LD, and stable disease (SD) as a decrease or increase less than PR or PD based on anatomic assessment. Patients with CR or PR will be defined as responders, whereas those with PD or SD are defined as non-responders.
Overall survival | up to 12 months
  The overall survival will be measured from the day of diagnosis to the date of death
Progression-free survival | up to 12 months
  The progression-free survival (PFS) will be measured from the day of diagnosis to the date of progressive disease.

IPD SHARING:
Plan to Share IPD: No